CLINICAL TRIAL: NCT06628817
Title: The Intensive Care Bundle with Mortality Reduction in Acute Ischemic Stroke Trial
Acronym: ICB-MRAIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Lou, Prof. Dr., Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ICB-MRAIS
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke
Keywords: quality improvement
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Hospitals assigned to the experimental group will receive a combined management intervention based on self-feedback from the online platform, including: a continuous automated medical quality monitoring and feedback system on the online platform, self-feedback and teamwork based on video conferencing, multidisciplinary online education, offline on-site supervision, and standardized intervention in the behavior of medical actors in the process of stroke treatment.
  Interventions: Radiation: The Intensive Care Bundle with Mortality Reduction
- No intervention (No Intervention): Hospitals in the control group only received self-feedback from the online platform in the neurology department, without receiving combined management intervention. / The neurology department of the control group hospitals only received self-feedback from the online platform, without receiving combined management intervention.

INTERVENTIONS:
Radiation: The Intensive Care Bundle with Mortality Reduction — a continuous automated medical quality monitoring and feedback system on the online platform, self-feedback and teamwork based on video conferencing, multidisciplinary online education, offline on-site supervision, and standardized intervention in the behavior of medical actors in the process of stroke treatment.
  Arms: Experimental Arm

SUMMARY:
Ischemic stroke, also known as cerebral infarction, accounts for as high as 60% to 80% of all stroke cases, and it is characterized by high morbidity, high disability rate, and high mortality rate. In recent years, acute ischemic stroke (AIS) has risen to the top of the list of causes of death in Chinese people, bringing a heavy burden on families, society and the country. In the process of continuous accumulation of evidence-based evidence, the management of stroke has gradually become systematic, and the demand for multi-disciplinary collaboration has become increasingly prominent, thus the concept of organized medical care has emerged.

Improving the prognosis of stroke faces multiple challenges, including timely identification of stroke patients, intravenous thrombolysis after clinical doctors evaluate indications and contraindications, reducing in-hospital stroke complications, accurately diagnosing the cause of stroke and implementing precise prevention. In the past, there were relatively few clinical trials on reducing mortality. The 2023 Dutch PRECIOUS study used metoclopramide, ceftriaxone and acetaminophen to prevent aspiration, infection and fever in elderly patients with acute stroke. The results showed that there was no significant difference in acute 90-day good functional outcomes and reduced mortality. The INTERACT3 trial results showed that for patients with acute cerebral hemorrhage, compared with conventional medical care, the use of a new combination management plan, namely early intensive blood pressure management, strict control of blood sugar elevation, body temperature control and anticoagulation therapy, can significantly reduce the risk of 6-month adverse functional prognosis in patients, improve the survival rate and quality of life of patients, and the possibility of patients being discharged within 7 days. Therefore, the use of a new combination management plan, including improving the efficiency of reperfusion therapy, reducing the occurrence of stroke complications, and carrying out precise etiological treatment, may reduce the mortality rate of patients.

The Zhejiang Stroke Online Platform can monitor the comprehensive information of treatment and management in the process of clinical doctors receiving AIS patients in real time. According to the self-feedback of each unit of the online platform, the provincial center conducts multi-level new combined management intervention on it. The purpose of this study is to explore whether the new combined management intervention measures can reduce the mortality rate of AIS patients on the basis of the implementation of stroke online platform monitoring.

DETAILED DESCRIPTION:
Ischemic stroke, also known as cerebral infarction, accounts for as high as 60% to 80% of all stroke cases, and it is characterized by high morbidity, high disability rate, and high mortality rate. In recent years, acute ischemic stroke (AIS) has risen to the top of the list of causes of death in Chinese people, bringing a heavy burden on families, society and the country. In the process of continuous accumulation of evidence-based evidence, the management of stroke has gradually become systematic, and the demand for multi-disciplinary collaboration has become increasingly prominent, thus the concept of organized medical care has emerged.

Improving the prognosis of stroke faces multiple challenges, including timely identification of stroke patients, intravenous thrombolysis after clinical doctors evaluate indications and contraindications, reducing in-hospital stroke complications, accurately diagnosing the cause of stroke and implementing precise prevention. In the past, there were relatively few clinical trials on reducing mortality. The 2023 Dutch PRECIOUS study used metoclopramide, ceftriaxone and acetaminophen to prevent aspiration, infection and fever in elderly patients with acute stroke. The results showed that there was no significant difference in acute 90-day good functional outcomes and reduced mortality. The INTERACT3 trial results showed that for patients with acute cerebral hemorrhage, compared with conventional medical care, the use of a new combination management plan, namely early intensive blood pressure management, strict control of blood sugar elevation, body temperature control and anticoagulation therapy, can significantly reduce the risk of 6-month adverse functional prognosis in patients, improve the survival rate and quality of life of patients, and the possibility of patients being discharged within 7 days. Therefore, the use of a new combination management plan, including improving the efficiency of reperfusion therapy, reducing the occurrence of stroke complications, and carrying out precise etiological treatment, may reduce the mortality rate of patients.

The Zhejiang Stroke Online Platform can monitor the comprehensive information of treatment and management in the process of clinical doctors receiving AIS patients in real time. According to the self-feedback of each unit of the online platform, the provincial center conducts multi-level new combined management intervention on it. The purpose of this study is to explore whether the new combined management intervention measures can reduce the mortality rate of AIS patients on the basis of the implementation of stroke online platform monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age of onset ≥ 18 years old;
2. AIS patients admitted to the hospital within 7 days of onset;
3. Obtain the informed consent of the patient or his/her family.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Modified rankin scale (mRS) scores of 4-6 at 1 year after acute stroke therapy | 1 year
  Modified rankin scale (mRS) scores of 4-6 at 1 year after acute stroke therapy